CLINICAL TRIAL: NCT05660798
Title: Effects of Switching From Cigarettes to Tobacco Heating System on Coronary Atherosclerosis Progression in Patients With Stable Coronary Artery Disease
Brief Title: Effects of Switching From Cigarettes to Tobacco Heating System on Coronary Atherosclerosis Progression
Acronym: SWITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: PMPSA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SWITCH01
Record Dates: First submitted 2022-10-12; First posted 2022-12-21 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Coronary Atherosclerosis; Nicotine Dependence
MeSH Terms: conditions — Coronary Artery Disease; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combustion tobacco (No Intervention)
- heated tobacco (Experimental)
  Interventions: Behavioral: heated tobacco - lifestyle intervention

INTERVENTIONS:
Behavioral: heated tobacco - lifestyle intervention — Patients unable (unwilling) to stop smoking will be randomized to either combustion (C) or heated (H) tobacco groups.
  Arms: heated tobacco

SUMMARY:
Objective:

To evaluate the impact of heated versus combustion tobacco products on progression of atherosclerosis in patients with CAD unable(unwilling) to quit smoking.

Rationale:

Despite the efforts to curb smoking and full awareness of its deleterious health impact, smoking remains a significant contributor to morbidity and mortality. Some health impact of smoking may be improved by other forms of cigarettes than traditional combustion, especially for subjects unwilling or unable to stop smoking. As recently as 2020, one of heated tobacco products (HTP)(IQOS) was FDA Authorized as a 'Reduced Exposure' product. The available evidence to date allows to conclude that the IQOS system heats tobacco but does not burn it, which significantly reduces the production of harmful and potentially harmful chemicals. Scientific studies have shown that switching completely from conventional cigarettes to the IQOS system significantly reduced body's exposure to harmful or potentially harmful chemicals. There is also evidence indicating lower levels of inflammatory markers and improved vascular function associated with use of heated tobacco products. However, it is unknown whether the reduction in the exposure translates into potential reduction of harm within cardiovascular system, as compared to the traditional (combustion) cigarettes.

The evidence is of crucial importance for patients with cardiovascular diseases, medical community, and national health authorities planning evidence based policies regarding HTP/cigarettes.

DETAILED DESCRIPTION:
Objective:

To evaluate the impact of heated versus combustion tobacco products on progression of atherosclerosis in patients with CAD unable(unwilling) to quit smoking.

Background Despite the efforts to curb smoking and full awareness of its deleterious health impact, smoking remains a significant contributor to morbidity and mortality. Some health impact of smoking may be improved by other forms of cigarettes than traditional combustion, especially for subjects unwilling or unable to stop smoking. As recently as 2020, one of heated tobacco products (HTP)(IQOS) was FDA Authorized as a 'Reduced Exposure' product. The available evidence to date allows to conclude that the IQOS system heats tobacco but does not burn it, which significantly reduces the production of harmful and potentially harmful chemicals. Scientific studies have shown that switching completely from conventional cigarettes to the IQOS system significantly reduced body's exposure to harmful or potentially harmful chemicals. There is also evidence indicating lower levels of inflammatory markers and improved vascular function associated with use of heated tobacco products. However, it is unknown whether the reduction in the exposure translates into potential reduction of harm within cardiovascular system, as compared to the traditional (combustion) cigarettes.

The evidence is of crucial importance for patients with cardiovascular diseases, medical community, and national health authorities planning evidence based policies regarding HTP/cigarettes.

Methods:

Prospective, single-centre, open-label, randomised study including 180 stable patients with coronary artery disease (CAD) as diagnosed on CCTA, without indications for invasive treatment, unable(unwilling) to quit smoking, randomised 1:1 to either heated (group H) or combustion (group C) tobacco products and followed for 18 months. The follow-up is accomplished with CCTA scan. The study clinical visits are planned at 1, 3, 6, 12, and 18 months.

The primary outcome is change in non calcified plaque volume at 18 months between H and C groups (intention to treat design).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged >18 years and <75 years
2. Subjects with stable chronic coronary syndrome defined as the presence of at least one coronary artery stenosis >=20% due to coronary plaque visible on coronary computed tomography angiography (CCTA), in an artery with a reference diameter > 2.0mm
3. History of smoking pack-years ≥10 (Pack-years will be calculated by taking the average number of cigarettes smoked per day divided by 20 and multiplied by the number of years smoked), based on self-reporting
4. Current smokers with a minimum of self-reported current smoking pattern of >10 cigarettes/day during the last 6 months prior to screening, smoking status will be verified based on a urinary cotinine test (cotinine ≥200 ng/mL)
5. Patients that have been advised to quit smoking and informed of a smoking risk and cessation programs (per local SOC) and who are still not willing to set a quit date within the next 30 days at screening
6. Stable treatment for coronary atherosclerosis according to the guidelines
7. Have understood the study and have signed informed consent

Exclusion Criteria:

1. Any acute cardiovascular event (i.e. ACS, MI, Stroke, TIA, Limb ischemia), unstable angina or revascularization within 30 days prior to screening
2. Planned coronary intervention (PCI, CABG) at screening
3. Previous CABG
4. Preexisting heart failure with reduced ejection fraction (EF <50%)
5. Severe uncontrolled hypertension (at the discretion of investigator)
6. Diabetes
7. Subjects with documented genetic familial hypercholesterolemia
8. Subjects have known serious infection or chronic inflammatory systemic disease (e.g. rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis)
9. Subjects have a known non-cardiovascular disease that is associated with poor prognosis (e.g. metastatic cancer)
10. Patient with currently active cancer or history of cancer within the last 5 years
11. Subjects have hypersensitivity or any other warnings listed in the local labeling for THS
12. Subjects have hypersensitivity to imaging iodine contrast agents
13. GFR<45 ml/min/1,73 m2
14. Subjects who could not participate for any reason other than medical (e.g., psychological and/or social reason) per Investigator's judgment
15. Subjects have any other clinical condition that would jeopardize the subject's safety while participating in this study, per Investigator's judgment
16. Female subject is pregnant or breast-feeding, or planning to become pregnant during the study
17. Subjects have previously participated in this study, or in an interventional study (drug or medical device) within 30 days of screening (participation in observational studies/registries allowed)
18. Subjects have a close affiliation with the investigational site: a close relative of the investigator, a person dependent on the investigational site (e.g. employee or student of the investigational site)
19. Subjects are current or former employee of the tobacco industry or their first-degree relatives (parent, child, spouse)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in non calcified plaque volume between H and C groups ("intention to treat") | 0-18 months
  CCTA based evaluation

SECONDARY OUTCOMES:
Change in total plaque volume | 0-18 months
  CCTA based evaluation
Change in plaque volume components (low attenuation, fibrous-fatty, fibrous, non-calcified plaque, calcified plaque) | 0-18 months
  CCTA based evaluation
Change in non calcified plaque volume between H and C groups ("as treated") | 0-18 months
  CCTA based evaluation
Change in lipid metabolism | 0-18 months
  Total cholesterol (TC) Triglycerides (TG) Lipoproteins: low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C) Apolipoproteins: apolipoprotein A1 (ApoA1), apolipoprotein B (ApoB) Lipoprotein(a) Lp(a)
Change in oxidative stress | 0-18 months
  8-Epi prostaglandin F2 alpha (8 epi PGF2α) Myeloperoxidase (MPO)
Change in inflammation | 0-18 months
  High-sensitivity C-reactive protein (hs CRP) White blood cell (WBC) counts Homocysteine Interleukins (IL-6) Fibrinogen
Change in platelet activation | 0-18 months
  11-dehydro-thromboxane B2 (11 DTX B2) Plasminogen activator inhibitor-1 (PAI-1) Tissue plasminogen activator (t-PA) Platelet count Mean platelet volume (MPV)
Change in endothelial dysfunction | 0-18 months
  P-selectin Metalloproteinase 9 (MMP-9)
Change in haemodynamic stress | 0-18 months
  N-terminal pro b-type natriuretic peptide (NT-proBNP)
Change in myocardial injury | 0-18 months
  high-sensitivity troponin T (hs-TnT)
Change in glycemia control | 0-18 months
  Fasting Blood Glucose, HbA1c
Change in physical activity | 0-18 months
  self reported, mobile device monitoring
Change in exposure to nicotine | 0-18 months
  4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol , Nicotine equivalents in spot urine , 2-cyanoethylmercapturic acid
SAFETY (ADVERSE OUTCOMES) | 0-18 months
  Independent DSMB will evaluate the outcomes
Change in self reported product use | 0-18 months
Change in quality of life | 0-18 months
  EQ5D-5L
Cost/effectiveness analysis | 0-18 months
Subgroup analysis (AGE/SEX/CO-MORBIDITIES) | 1-18 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biondi-Zoccai G, Sciarretta S, Bullen C, Nocella C, Violi F, Loffredo L, Pignatelli P, Perri L, Peruzzi M, Marullo AGM, De Falco E, Chimenti I, Cammisotto V, Valenti V, Coluzzi F, Cavarretta E, Carrizzo A, Prati F, Carnevale R, Frati G. Acute Effects of Heat-Not-Burn, Electronic Vaping, and Traditional Tobacco Combustion Cigarettes: The Sapienza University of Rome-Vascular Assessment of Proatherosclerotic Effects of Smoking ( SUR - VAPES ) 2 Randomized Trial. J Am Heart Assoc. 2019 Mar 19;8(6):e010455. doi: 10.1161/JAHA.118.010455. PMID 30879375
- [Background] Ikonomidis I, Vlastos D, Kostelli G, Kourea K, Katogiannis K, Tsoumani M, Parissis J, Andreadou I, Alexopoulos D. Differential effects of heat-not-burn and conventional cigarettes on coronary flow, myocardial and vascular function. Sci Rep. 2021 Jun 3;11(1):11808. doi: 10.1038/s41598-021-91245-9. PMID 34083663